CLINICAL TRIAL: NCT01912950
Title: Randomized, Controlled, Open-Label Pilot Study of a Novel IPL for Removal of Unwanted Fine Hair
Brief Title: Pilot Study of a Novel IPL for Removal of Unwanted Fine Body Hair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cutera Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-13-PW01
Record Dates: First submitted 2013-07-18; First posted 2013-07-31 (Estimated); Results first posted 2023-02-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-01

CONDITIONS: Hypertrichosis
Keywords: intense pulsed light; IPL; healthy volunteer; light-based hair removal; hair removal; epilation; laser hair removal; permanent hair reduction
MeSH Terms: conditions — Hypertrichosis | interventions — Intense Pulsed Light Therapy; Hair Removal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prowave LX IPL (Experimental): One area on forearm will receive treatment with Prowave LX IPL
  Interventions: Device: Prowave LX IPL
- No Treatment (No Intervention): No treatment administered on one area of forearm

INTERVENTIONS:
Device: Prowave LX IPL
  Other Names: Prowave; Prowave LX; Cutera Prowave LX; Intense Pulsed Light; IPL; Flashlamp Infared device; Hair removal
  Arms: Prowave LX IPL

SUMMARY:
The purpose of this randomized, controlled, open-label pilot study is to evaluate the safety and efficacy of a novel intense pulsed light (IPL) device for removal of unwanted fine body hair.

Subjects will have IPL treatment on one forearm area. Another area will serve as the un-treated control area. Subjects will be followed at 12-weeks post-final treatment.

ELIGIBILITY:
Inclusion Criteria:

* Female or Male, 18 to 65 years of age (inclusive).
* Fitzpatrick Skin Type I - III.
* Subject has black or dark brown unwanted arm hair of fine texture.
* Willing to have the hair removal procedure on one forearm only, and within the designated study treatment area.
* Willing and able to adhere to the treatment and follow-up schedule, and the study "Before and After Procedure Instructions".
* Willing to refrain from shaving the treatment area for 5 days prior to each study visit.
* Must be able to read, understand and sign the Informed Consent Form.
* Must agree not to use hair removal products, such as topical chemical depilatories, or undergo any other hair removal procedure during the study, such as other laser and light therapies or waxing.
* Willing to refrain from excess sun exposure and willing to wear sunscreen on the treatment area during the study (including the follow-up period).
* Willing to have digital photographs taken of the treatment area and agree to use of photographs for presentation, educational or marketing purposes.
* Must be in good health, as determined by the Investigator.
* Must be post-menopausal or surgically sterilized, or using a medically acceptable form of birth control at least 3 months prior to enrollment and during the entire course of the study.

Exclusion Criteria:

* Participation in a clinical trial of another device or drug within 6 months prior to enrollment, or during the study.
* Had any type of professional hair removal procedure, such as laser, light-based, RF or electrolysis, in the treatment area within 12 months of study participation.
* Had other epilation treatment, such as waxing or mechanical epilator, in the treatment area within 6 months of study participation.
* Subject shows signs of actinic bronzing or recent tanning in the treatment area, and unable/unlikely to refrain from tanning during the study.
* Subject is pregnant and/or breastfeeding.
* Suffering from significant concurrent illness, such as diabetes mellitus or pertinent neurological disorders.
* Having malignant or pre-malignant lesions in the treatment area, or history of a malignant skin disease.
* Current acute or chronic skin infections or inflammatory processes, affecting the treatment area, such as dermatitis.
* Currently using immunosuppressive medications or history of immunosuppression/immune deficiency disorder, such as psoriasis, eczema, vitiligo, systemic lupus erythematosus or scleroderma.
* Current use of any medication that is known to increase sensitivity to light, such as tetracycline.
* Currently undergoing systemic chemotherapy or radiation treatment for cancer, or history of treatment within 3 months of study participation.
* Suffering from coagulation disorders or taking prescription anticoagulation medications.
* History of keloid formation, hypertrophic scarring or abnormal/delayed wound healing.
* History of seizure disorders due to light.
* History of diseases stimulated by heat, such as recurrent herpes zoster in the treatment area, unless treatment is conducted following a prophylactic regimen.
* History of pigmentary disorders, particularly tendency for hyper- or hypo-pigmentation.
* History of tattoo, permanent make-up or semi-permanent or permanent tissue fillers in the treatment area.
* Systemic use of a retinoid (such as Accutane) or corticosteroid within 6 months of study participation.
* Current smoker or history of smoking within 12 months of study participation.
* Anytime in life, had used gold therapy (gold salts) for disorders such as rheumatologic disease or lupus.
* As per the Investigator's discretion, any physical or mental condition which might make it unsafe for the subject to participate in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2013-12; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neil Sadick, Principal Investigator — Study Principal Investigator
Locations (1):
- Sadick Research Group, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: areas on the forearm
Groups:
- All Study Participants: Each subject will receive hair removal treatments with the Prowave LX IPL. Each subject will have one designated treatment area on the foreman and one un-treated control area.
Period: Overall Study
Arm/Group | All Study Participants
Started | 11; 22 areas on the forearm
Treated Areas on the Forearm | 11; 11 areas on the forearm
Untreated Areas on the Forearm | 11; 11 areas on the forearm
Completed | 7; 14 areas on the forearm
Not Completed | 4; 8 areas on the forearm

BASELINE CHARACTERISTICS:
Groups:
- All Enrolled Subjects: All enrolled subjects receiving treatment
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Percent Hair Reduction Between Treatment Arm and Non-treated Control Arm at 12 Weeks Post Final Treatment
Time Frame: 12-weeks
Measure: Mean (Full Range); unit: percent reduction
Groups:
- Prowave LX IPL: Treatment with Prowave LX IPL
- No Treatment: No treatment administered
Arm/Group | Prowave LX IPL | No Treatment
Number analyzed (Participants) | 7 | 7
percent reduction | 41 [-62 to 97] | 27 [-60 to 85]

ADVERSE EVENTS:
Time Frame: 12 weeks
Groups:
- Prowave LX IPL: Prowave LX IPL on one area of the forearm
Arm/Group | Prowave LX IPL | No Treatment
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 5/11 | 0/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Prowave LX IPL (N=11) | No Treatment (N=11)
Erythema (Skin and subcutaneous tissue disorders) | 5 | 0
Edema (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No